CLINICAL TRIAL: NCT01523054
Title: A Pharmacokinetic and Pharmacodynamic Study Comparing Metoprolol IR and Metoprolol CR/XL Subsequent to Initial Treatment With Intravenous and/or Oral Metoprolol in Patients With Suspected Acut Myocardial Infarction
Brief Title: Metoprolol in Acute Myocardial Infarction. A PK/PD Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SH-MET-0027
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Acute Myocardial Infarction
Keywords: metoprolol, acute myocardial infarction, pharmacokinetics, pharmacodynamics
MeSH Terms: interventions — Metoprolol

ARMS (2):
- Metoprolol- Toprol XL (Experimental): Metoprolol extended release (CR/XL) tablet 200 mg once daily
  Interventions: Drug: Metoprolol- Toprol XL
- Metoprolol- Lopressor (Active Comparator): Metoprolol immediate release (IR) tablet
  Interventions: Drug: Metoprolol- Lopressor

INTERVENTIONS:
Drug: Metoprolol- Toprol XL — Extended release tablet, 200mg once daily for 4 days
  Arms: Metoprolol- Toprol XL
Drug: Metoprolol- Lopressor — Immediate release tablet, Day 1 50 mg four times daily, Day 2, 3 and 4 100 mg twice daily
  Arms: Metoprolol- Lopressor

SUMMARY:
The objective of the study was to compare treatment with two different oral formulations of metoprolol, metoprolol immediate release (IR) and metoprolol extended release (CR/XL) in patients with acute myocardial infarction regarding the following:

Pharmacokinetics, peak and trough plasma concentrations and area under the plasma concentration curve.

Pharmacodynamics, hourly means of Holter recorded heart rate. Tolerability. An open, randomised design with two parallel groups was employed.

DETAILED DESCRIPTION:
A pharmacokinetic and pharmacodynamic study comparing metoprolol IR and metoprolol CR/XL subsequent to initial treatment with intravenous and/or oral metoprolol in patients with suspected acut myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients admitted to the CCU with suspected acute myocardial infarction
* Age 18 years or older
* Treated with and tolerated the full dose of metoprolol IR 50 mr four times daily or metoprolol CR/XL 200 mg once daily on study day 1
* Expected to stay in the CCU until the morning of study day 4
* Sinus rhythm on the day of admission and at randomisation

Exclusion Criteria:

* Pregnancy or childbearing potential without adequate contraception
* Participation in a clinical study during the last 30 days or previous randomisation in the present study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2000-02; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile in terms of Cmax, Cmin, AUC | Treatment duration: 4 days
  Assesment following multiple dosing of metoprolol CR/XL 200 mg once daily, or multiple dosing of metoprolol IR 200 mg daily in divided doses
Pharmacodynamics in terms of Hourly means of heart rate (Holter recorded) | Treatment duration: 4 days
  Assesment following multiple dosing of metoprolol CR/XL 200 mg once daily, or multiple dosing of metoprolol IR 200 mg daily in divided doses
Safety profile in terms of adverse events | Treatment duration: 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Dag Elmfeldt, MD, PHD, Study Director — AstraZeneca R&D Mölndal